CLINICAL TRIAL: NCT04993105
Title: Effects of Graston Assisted Soft Tissue Mobilization in Patients With Chronic Plantar Fasciitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00869 Maham Nasir
Record Dates: First submitted 2021-06-11; First posted 2021-08-06 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Plantar Fascitis
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: study will evaluate the effects of Graston assisted soft tissue mobilization on the patients with plantar fasciitis .Study will include two groups , one will be treated with graston and one will be treated without graston in the time period of two weeks.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- B (exercise + graston): (Experimental): In graston + exercises treatment will be same but after exercises added with proper application of graston which included application of a cream to the posterior calf and plantar foot from the knee to the toes to reduce friction on the skin.The Graston tools will be then used to mobilize the tissues of the triceps surf and plantar foot. In areas of increased tissue restriction, more aggressive pressure with graston was applied using increased force and shorter strokes over the areas of restriction was offered as needed for pain management after each session. This will be continued for three sessions. NPRS score, score on FADI and dorsiflexors range will be assessed after treatment of two weeks. Along with conventional treatment.
  .
  Interventions: Other: Exercise + Graston.
- A (exercise only) (Active Comparator): Exercises only. Patients will be given gastrocnemius stretching, plantar fascia stretching, myofascial release and then graston will be given as sham treatment for 10 minutes after applying cream (applying graston on skin but not giving enough pressure).
  Interventions: Other: exercise only

INTERVENTIONS:
Other: Exercise + Graston. — In graston + exercises treatment will be same but after exercises added with proper application of graston which included application of a cream to the posterior calf and plantar foot from the knee to the toes to reduce friction on the skin.The Graston tools will be then used to mobilize the tissues of the triceps surae and plantar foot. In areas of increased tissue restriction, more aggressive pressure with graston was applied using increased force and shorter strokes over the areas of restrictionIce was offered as needed for pain management after each session. This will be continued for three sessions. NPRS score, score on FADI and dorsiflexors range will be assessed after treatment of two weeks. Along with conventional treatment.
  .
  Other Names: exercise only
  Arms: B (exercise + graston):
Other: exercise only — gastrocnemius and plantarstretching
  Arms: A (exercise only)

SUMMARY:
study was conducted to check the effectiveness of graston on patients with chronic plantar fasciitis. After screening from inclusion exclusion criteria.Data will be randomly divided in two groups.

Graston assisted release of plantar fascia is used for soft tissue mobilization. Pain level using NPRS, score on FADI and dorsiflexion restriction using LUNGE test will be performed before any treatment.

DETAILED DESCRIPTION:
Plantar fasciitis is one of the most common cause of pain in foot and calf areas effecting up to 10% of the total population.(1) On assessment of such patients pain on calcaneal tuberosity on passive dorsiflexion is very common.(2) Common features include sharp stabbing pain specially in morning which subsides after brief walking but may return after prolong period of weight bearing and walking.In general, plantar fasciitis occurs when the plantar fascia is injured from too much pressure or activity, but there is often not a clear cause or triggering event(3)People who are overweight and people who have tight calf muscles, high-arched feet, or flat feet are at risk of plantar fasciitis(4).

Simple measures can often be taken to lessen the symptoms of plantar fasciitis(5). If a clear cause such as a sudden increase in high-impact exercise can be identified, then decreasing the amount of physical activity may be helpful.(6)Daily stretching of the plantar fascia and the calf muscles should be performed, and ice can be applied to the affected area for 10 to 20 minutes at a time 2 to 3 times per day. Wearing shoes with good arch supports can also improve symptoms, and taping the bottom of the feet or using shoe inserts called orthotics are other ways to provide additional foot support. .(6) Over-the-counter anti-inflammatory medications such as ibuprofen may provide short-term relief(7). If pain persists, steroid injections may be given into the foot to reduce the pain. Although most people experience improvement or resolution of symptoms over time, surgery may be considered in rare cases if the pain does not improve after several months of conservative treatments(8). Graston is a used for soft tissue mobilization. Graston Technique is performed by specifically designed stainless steel instruments with beveled edges to perform soft tissue mobilization graston is used in a multi direction strokes on skin at a 30° to 60° angle to the treatment site(8)This technique allows the clinician to feel irregularities in the soft tissue texture through the movement of the gliding tools(8)In addition to removing scar tissue adhesions, Graston instruments have been applied to boost the proliferation of extracellular matrix fibroblasts, improve ion transport, and decrease cell matrix adhesions as has been hypothesized with transverse frictional massage and extra corporeal shock wave therapy.(6)Studies have shown that the controlled micro trauma induced through GT increased fibroblasts recruitment and activation in an animal model. Additional studies have shown clinical efficacy using GT for the treatment of carpal tunnel syndrome, lumbar compartment syndrome(7) and trigger thumb(8). Graston instrument has been used for relieving pressure of soft tissue mobilization and release very effectively for years. It is used by manual therapist and is also known as instrument assisted soft tissue mobilization(IASTM). The instruments are specially designed for manual therapist to identify the areas of adhesion in soft tissue and focus on the release.As proved by Carey-Loghmani and Hammer the GISTM is used to detect and treat soft tissue lesions.The application of the GISTM initiates the inflammatory process, which allows for healing and scar tissue remodeling to take place(9). Although a recent systematic review have reported on current evidence to support the use of conservative interventions for individuals identified as having CPHP. Martin et al reported that soft-tissue mobilization procedures should also be considered in the plan of care for individuals with CPHP(10).

Recent research suggests that plantar "fasciitis" manifests itself as a noninflammatory degenerative process, and hence, the term fasciosis may be more appropriate.(6) Brian looney et al proved graston to be an effective tool to increase pain and dorsiflexion range in patients with plantar fasciitis through case series(11). The authors reported that the participants demonstrated clinically meaningful improvements in pain ratings and functional improvements in Global Rating of Change Scale and Lower Extremity Functional Scale scores(11)Daniels and Morrell reported the effectiveness of using the Graston technique to perform IASTM in addition to joint manipulation to manage a 10-year-old male athlete with bilateral plantar fasciitis(12). In addition, the biologic evidence that suggests that PF is not truly an inflammatory condition but one of fibrosis supports the theorized mechanism behind the graston(2) .Perhaps the use of instruments allows the clinician to introduce a more controlled amount of micro trauma into an area of scar tissue or excessive fibrosis(8). Research suggests that the response of this microtrauma would result in the healing process by initiating inflammatory phase of healing and, ultimately, tissue remodeling through proper realignment of collagen fibers(11).A pilot study by Edward R. Jones et al demonstrates that inclusion of IASTM using the Graston technique for chronic plantar heel pain lasting longer than 6 weeks is a feasible intervention warranting further study(13). Andrew L. Miners and Tracy L. Bougie showed a specific protocol of heat, graston assisted soft tissue mobilization, eccentric exercise, stretching, and cryotherapy appeared to facilitate a rapid and complete recovery from chronic Achilles tendinopathy(14).

ELIGIBILITY:
Inclusion Criteria:

The study includes patients from the age group of 35 to 50 years.

* The study includes patients with plantar heel pain from more than 6 weeks
* The study includes patients with restricted dorsiflexion which will be measured by lunge's test
* Pain in morning (decrease with activity)

Exclusion Criteria:

* The study acute patient with plantar pain.
* No history of serious underlying pathology, nerve root compromise, structural deformities, genetic spinal disorders or previous spinal surgery

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
effects of graston on pain in patients with plantar fasciitis. | 6 months
  Pain will be evaluated by NPRS on scale of to 10

SECONDARY OUTCOMES:
effects of graston on range of motion in patients with plantar fasciitis. | 6 months
  Range of motion will be calculated by Lunge test.
effects of graston assisted soft tissue mobilization on Foot and ankle function and disability. | 6 months
  Will be calculated by Foot and ankle disability Index.

CONTACTS AND LOCATIONS:
Overall Officials: Lal Gul Khan, MScPT, Principal Investigator — Riphah International University
Locations (1):
- Rawal General and Dental Hospital, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roxas M. Plantar fasciitis: diagnosis and therapeutic considerations. Altern Med Rev. 2005 Jun;10(2):83-93. PMID 15989378
- [Background] Aldridge T. Diagnosing heel pain in adults. Am Fam Physician. 2004 Jul 15;70(2):332-8. PMID 15291091
- [Background] Atkins D, Crawford F, Edwards J, Lambert M. A systematic review of treatments for the painful heel. Rheumatology (Oxford). 1999 Oct;38(10):968-73. doi: 10.1093/rheumatology/38.10.968. PMID 10534547
- [Background] DiGiovanni BF, Nawoczenski DA, Lintal ME, Moore EA, Murray JC, Wilding GE, Baumhauer JF. Tissue-specific plantar fascia-stretching exercise enhances outcomes in patients with chronic heel pain. A prospective, randomized study. J Bone Joint Surg Am. 2003 Jul;85(7):1270-7. doi: 10.2106/00004623-200307000-00013. PMID 12851352
- [Background] Lemont H, Ammirati KM, Usen N. Plantar fasciitis: a degenerative process (fasciosis) without inflammation. J Am Podiatr Med Assoc. 2003 May-Jun;93(3):234-7. doi: 10.7547/87507315-93-3-234. PMID 12756315
- [Background] Muth CC. Plantar Fasciitis. JAMA. 2017 Jul 25;318(4):400. doi: 10.1001/jama.2017.5806. No abstract available. PMID 28742914
- [Background] Hammer WI, Pfefer MT. Treatment of a case of subacute lumbar compartment syndrome using the Graston technique. J Manipulative Physiol Ther. 2005 Mar-Apr;28(3):199-204. doi: 10.1016/j.jmpt.2005.02.010. PMID 15855909
- [Background] Howitt S, Wong J, Zabukovec S. The conservative treatment of Trigger thumb using Graston Techniques and Active Release Techniques. J Can Chiropr Assoc. 2006 Dec;50(4):249-54. PMID 17549185
- [Background] Martin RL, Davenport TE, Reischl SF, McPoil TG, Matheson JW, Wukich DK, McDonough CM; American Physical Therapy Association. Heel pain-plantar fasciitis: revision 2014. J Orthop Sports Phys Ther. 2014 Nov;44(11):A1-33. doi: 10.2519/jospt.2014.0303. PMID 25361863
- [Background] Looney B, Srokose T, Fernandez-de-las-Penas C, Cleland JA. Graston instrument soft tissue mobilization and home stretching for the management of plantar heel pain: a case series. J Manipulative Physiol Ther. 2011 Feb;34(2):138-42. doi: 10.1016/j.jmpt.2010.12.003. PMID 21334547
- [Background] Daniels CJ, Morrell AP. Chiropractic management of pediatric plantar fasciitis: a case report. J Chiropr Med. 2012 Mar;11(1):58-63. doi: 10.1016/j.jcm.2011.06.009. PMID 22942843
- [Background] Jones ER, Finley MA, Fruth SJ, McPoil TG. Instrument-Assisted Soft-Tissue Mobilization for the Management of Chronic Plantar Heel Pain: A Pilot Study. J Am Podiatr Med Assoc. 2019 May;109(3):193-200. doi: 10.7547/16-105. Epub 2019 Mar 27. PMID 30916579
- [Background] Miners AL, Bougie TL. Chronic Achilles tendinopathy: a case study of treatment incorporating active and passive tissue warm-up, Graston Technique, ART, eccentric exercise, and cryotherapy. J Can Chiropr Assoc. 2011 Dec;55(4):269-79. PMID 22131563
- [Background] Young IA PT, DSc, Dunning J PT, DPT, Butts R PT, PhD, Mourad F PT, DPT, Cleland JA PT, PhD. Reliability, construct validity, and responsiveness of the neck disability index and numeric pain rating scale in patients with mechanical neck pain without upper extremity symptoms. Physiother Theory Pract. 2019 Dec;35(12):1328-1335. doi: 10.1080/09593985.2018.1471763. Epub 2018 Jun 1. PMID 29856244